CLINICAL TRIAL: NCT04940910
Title: A 8 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Black Rice Bran Extract on Immune Enhancement
Brief Title: The Efficacy and Safety of Black Rice Bran Extract on Immune Enhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JARM-IE-BRBE
Record Dates: First submitted 2021-06-07; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Immunity
Keywords: Black Rice Bran; Immunity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black rice bran extract group (Experimental): 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal(1.52 g/day, Black rice bran extract 1 g/day)
  Interventions: Dietary Supplement: Black rice bran extract
- Placebo group (Placebo Comparator): 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal(1.52 g/day, Black rice bran extract 0 g/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Black rice bran extract — 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal, for 8 week
  Arms: Black rice bran extract group
Dietary Supplement: Placebo — 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal, for 8 week
  Arms: Placebo group

SUMMARY:
This study was conducted to investigate the efficacy and safety of Black rice bran extract on immune enhancement.

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Black rice bran extract on immune enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 19 and under 75 years
* After fully hearing and fully understanding this clinical trials, those who agree to voluntarily decide to participate and to comply with the notice

Exclusion Criteria:

* If screening shows that the white blood cell(WBC) is less than 3000/㎕ or more than 8000/㎕
* Those who received influenza vaccination within 3 months before first intake of intervention
* Those who have a body mass index(BMI) of less than 18.5 kg / m^2 or greater than 35 kg / m^2 at the screening
* Those who have a clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry, musculoskeletal system, inflammatory and hematologic and gastrointestinal disorders
* Those who take a medication or health function food that affects your promotion of immunity within 1 month prior to the screening
* Those who have received antipsychotic medication within 3 months before screening
* Those who alcoholic or drug abuse suspected
* Those who participated in other clinical trials within 3 months before screening
* Laboratory test by show the following results

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Those who doesn't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
Changes of Natural Killer cell activity | baseline and 8 weeks
  Natural Killer cell activity was measured in study baseline and 8 week. A ratio of effector cell and target cell was 2.5:1, 5:1, 10:1.
  (Experimental - Effector Spontaneous - Target Spontaneous) / (Target Maximum - Target Spontaneous) × 100

SECONDARY OUTCOMES:
Changes of Interleukin-2, Interleukin-12, Interferon-Gamma and Tumor necrosis factor-alpha | baseline and 8 weeks
  For blood Interleukin-2, Interleukin-12, Interferon-Gamma and Tumor necrosis factor-alpha analysis, collect 3 ml of blood in one serum separate tube for 5 ml, leave at room temperature for 30 minutes for clotting, after then centrifuge at 3000 rpm (or 2000 xg) for 10 minutes.
Changes of Wisconsin Upper Respiratory Symptom Survey-21(WURSS-21) | baseline, 4 weeks and 8 weeks
  The Wisconsin Upper Respiratory Symptom Survey-21 will investigate on the day of visit (1st, 2nd and 3rd visits).
  The Wisconsin Upper Respiratory Symptom Survey-21 consists of seven stages, including individual symptoms, functional quality of life, and overall improvement. Find the total score of symptoms by obtaining the sum of symptom questions, and the total score of quality of life by obtaining the sum of life questions. Additionally, the sum of the total points of symptoms and quality of life is obtained.
  * All items of symptom score rank on a seven-point scale(1=very mild and 7=severe), where a higher score means higher severity. The symptom score ranges from 0(Do not have this symptom) to 70.
  * All items of quality of life score rank on a seven-point scale(1=very mildly and 7=severely), where a higher score means higher severity. The quality of life score ranges from 0(Not at all) to 63.
  * Therefore, the total score ranges from 0 to 133.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea